CLINICAL TRIAL: NCT05890456
Title: Efficacy of the Students With Involved Families and Teachers (SWIFT) Program for Students With Emotional and Behavioral Disorders
Brief Title: Students With Involved Families and Teachers
Acronym: SWIFT-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Responsible Party: Principal Investigator, Rohanna Buchanan, Research Scientist, Oregon Social Learning Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R324A190122
Record Dates: First submitted 2023-02-22; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Emotional Regulation; Adolescent Behavior; Parenting
Keywords: Positive Parenting; Behavior Regulation; Academic Success
MeSH Terms: conditions — Emotional Regulation; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Students and their families will be randomly assigned to the SWIFT Program or SAU conditions. A blocked design will be used where randomization will occur at the individual level within each school once a family has agreed to study participation. This way variation between schools (blocks) will not affect the standard errors of treatment effect estimates. Key outcomes will be tested at Time 1 (T1, baseline), Time 2 (T2, 6 months post-baseline), Time 3 (T3, 12 months post-baseline), and Time 4 (T4, 18 months post-baseline).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): The SWIFT Program is a 9-12 month intervention that includes four components: (a) behavioral progress monitoring, (b) clinical supervision of the intervention elements and coordination with the school, (c) parent support to promote parent engagement/collaboration with the school and study routines in the home, and (d) behavioral skills coaching for students. SWIFT students will continue to receive any school-based services that were receiving prior to entering the study.
  Interventions: Behavioral: Students with Involved Families and Teacher Program
- Services As Usual Control (Active Comparator): The SAU students and families will continue to receive any services that they were receiving prior to their entry into the study. These may include school-based interventions and supports and related services as required in the student's Individualized Education Program.
  Interventions: Behavioral: Services As Usual

INTERVENTIONS:
Behavioral: Students with Involved Families and Teacher Program — The SWIFT Program is a 9-12 month intervention that includes four components: (a) behavioral progress monitoring, (b) clinical supervision of the intervention elements and coordination with the school, (c) parent support to promote parent engagement/collaboration with the school and study routines in the home, and (d) behavioral skills coaching for students.
  Other Names: SWIFT
  Arms: Treatment Arm
Behavioral: Services As Usual — The SAU students and families will continue to receive any services that they were receiving prior to their entry into the study. These may include school-based interventions and supports and related services as required in the student's Individualized Education Program.
  Other Names: SAU
  Arms: Services As Usual Control

SUMMARY:
PURPOSE: In the proposed project, the investigators seek to examine whether the SWIFT Program might be efficacious to improve students' prosocial skills and emotion and behavior regulation and improve home-school communication and the use of positive parenting practices for families. The investigators will also test whether the SWIFT program might be efficacious to improve students' longer-term school adjustment and parents' involvement in school.

SETTING: Study activities will take place in ten school districts in Lane County, OR. The districts have approximately 10,000 middle school students (Grades 6-8), and approximately 60% of students are eligible for free and reduced price lunch. Some participating districts participated in the IES-funded Goal 2 study to develop the SWIFT Program.

POPULATION: 320 students in Grades 6-8 who are receiving special education services for emotional or behavioral disorders, and transitioning or at risk of transitioning between school settings and placements will be recruited. Parents and content area teachers of all participating students will be recruited to complete assessment measures. It is expected that up to 15% of the children in the study will be of Latino ethnicity and approximately 60% will be European-American and 10-20% will be of other or multiple ethnicities.

INTERVENTION: The SWIFT Program is a 9-12 month intervention that includes four components: (a) behavioral progress monitoring, (b) case management of the intervention elements and coordination with the school, (c) parent support to promote parent engagement/collaboration with the school and study routines in the home, and (d) behavioral skills coaching for students.

SERVICES AS USUAL (SAU) CONTROL CONDITION: The SAU students and families will continue to receive any services that they were receiving prior to their entry into the study (as will the SWIFT students and families). These may include school-based interventions and supports and related services as required in the student's IEP.

ELIGIBILITY:
Inclusion Criteria:

* Students in grades 5 through 8
* In school districts in the the Lane Education Service District
* Eligible for or at risk of eligibility for special education services for emotional or behavior disorders
* Transitioning or at risk of transitioning between school settings or placements
* English or Spanish speaking

Exclusion Criteria:

* Students receiving intensive family and school support services from local community mental health agencies
* Students with a hearing or vision impairment that would limit participation in the program components or the assessment protocol.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean Changes in Youth Emotional and Behavioral Outcomes from Baseline to 6 Months Post-Baseline | Baseline to 6 Months Post-Baseline
  Emotion regulation skills measured by the Emotion Regulation Checklist. Measured at Baseline and 6 months post-Baseline.
Mean Changes in Youth Emotional and Behavioral Outcomes from Baseline to 6 Months Post-Baseline | Baseline to 6 Months Post-Baseline
  Psychopathological behaviors measured by the Child Behavior Checklist. Measured at Baseline and 6 months post-Baseline.
Mean Changes in Youth Academic Outcomes from Baseline to 6 Months Post-Baseline | Baseline to 6 Months Post-Baseline
  Academic outcomes measured by youth grades. Measured at Baseline and 6 months post-Baseline.
Mean Changes in Youth Academic Outcomes from Baseline to 6 Months Post-Baseline | Baseline to 6 Months Post-Baseline
  Academic outcomes measured by EasyCBM score. Measured at Baseline and 6 months post-Baseline.
Mean Changes in Parenting Outcomes from Baseline to 6 Months Post-Baseline | Baseline to 6 Months Post-Baseline
  Parenting outcomes measured by the Parenting Practices Questionnaire. Measured at Baseline and 6 months post-Baseline.

SECONDARY OUTCOMES:
Stability in School Placement from Baseline to 6 Months | Baseline to 6 Months Post-Baseline
  Measured by number of school placement moves. Measured at Baseline and 6 months post-Baseline.
Mean Changes in Youth Emotional and Behavioral Outcomes from Baseline to 12 Months | Baseline to 12 Months Post-Baseline
  Emotion regulation skills measured by the Emotion Regulation Checklist. Measured at Baseline and 12 months post-Baseline.
Mean Changes in Youth Emotional and Behavioral Outcomes from Baseline to 12 Months | Baseline to 12 Months Post-Baseline
  Psychopathological behaviors measured by the Child Behavior Checklist. Measured at Baseline and 12 months post-Baseline.
Mean Changes in Youth Academic Outcomes from Baseline to 12 Months Post-Baseline | Baseline to 12 Months Post-Baseline
  Academic outcomes measured by youth grades. Measured at Baseline and 12 months post-Baseline.
Mean Changes in Youth Academic Outcomes from Baseline to 12 Months Post-Baseline | Baseline to 12 Months Post-Baseline
  Academic outcomes measured by EasyCBM score. Measured at Baseline and 12 months post-Baseline.
Mean Changes in Parenting Outcomes from Baseline to 12 Months Post-Baseline | Baseline to 12 Months Post-Baseline
  Parenting outcomes measured by the Parenting Practices Questionnaire. Measured at Baseline and 12 months post-Baseline.
Stability in School Placement from Baseline to 12 Months | Baseline to 12 Months Post-Baseline
  Measured by number of school placement moves. Measured at Baseline and 12 months post-Baseline.
Mean Changes in Youth Emotional and Behavioral Outcomes from Baseline to 18 Months | Baseline to 18 Months Post-Baseline
  Psychopathological behaviors measured by the Child Behavior Checklist. Measured at Baseline and 18 months post-Baseline.
Mean Changes in Youth Emotional and Behavioral Outcomes from Baseline to 18 Months | Baseline to 18 Months Post-Baseline
  Emotion regulation skills measured by the Emotion Regulation Checklist. Measured at Baseline and 18 months post-Baseline.
Mean Changes in Youth Academic Outcomes from Baseline to 18 Months Post-Baseline | Baseline to 18 Months Post-Baseline
  Academic outcomes measured by youth grades. Measured at Baseline and 18 months post-Baseline.
Mean Changes in Youth Academic Outcomes from Baseline to 18 Months Post-Baseline | Baseline to 18 Months Post-Baseline
  Academic outcomes measured by EasyCBM score. Measured at Baseline and 18 months post-Baseline.
Mean Changes in Parenting Outcomes from Baseline to 18 Months Post-Baseline | Baseline to 18 Months Post-Baseline
  Parenting outcomes measured by the Parenting Practices Questionnaire. Measured at Baseline and 18 months post-Baseline.
Stability in School Placement from Baseline to 18 Months | Baseline to 18 Months Post-Baseline
  Measured by number of school placement moves. Measured at Baseline and 18 months post-Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Rohanna Buchanan, PhD, Principal Investigator — Oregon Social Learning Center
Locations (1):
- Oregon Social Learning Center, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Per IES requirements...